CLINICAL TRIAL: NCT04002492
Title: Effects of a Weight Based Training Program on Bone Density, Cognition, and Quality of Life of Multiple Sclerosis Patients
Brief Title: Effects of a Weight Based Training Program on MS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Holy Name Medical Center, Inc. (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Mary Ann Picone, MD, Medical Director of Holy Name Comprehensive Care Center, Holy Name Medical Center, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: US-MSG-17-11209
Record Dates: First submitted 2019-06-14; First posted 2019-06-28 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
Keywords: sarcopenia; osteopenia; exercise; body weight training; bone density; demyelination; cognition
MeSH Terms: conditions — Multiple Sclerosis; Sarcopenia; Bone Diseases, Metabolic; Motor Activity; Demyelinating Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Addition of bodyweight training (Experimental): All participants in this study fall into this non randomized single group. These participants will complete a total of 12 bodyweight training sessions over a six to eight week time period. Participants will attend one session per week at Holy Name Medical Center's Physical Therapy Center and will train for one session at their home or chosen location with the aid of a video guide.
  Interventions: Behavioral: Bodyweight training

INTERVENTIONS:
Behavioral: Bodyweight training — Video guided and physical therapist guided bodyweight training sessions will be performed twice a week for 6 (to 8) weeks. These sessions include the following five workouts at 3 sets of 10 repetitions: step ups, calf raises, wall push ups, chair squats, and chair dips.

SUMMARY:
Low bone density is a health risk in older adults and especially people with multiple sclerosis (MS) due to steroid treatments and less mobility. Bone density is a measurement of how dense or strong bones are. Weight-based training may be one method in strengthening bones and providing a beneficial treatment for MS patient rehabilitation. Weight based training involves performing exercises without the use of actual weights, and instead with one's own bodyweight. This study aims to look at the effects of weight-based training on bone density, cognition (ability to learn and understand), and other quality of life issues (i.e. depression) in MS patients.

DETAILED DESCRIPTION:
This study aims to observe if there is a correlation between increasing one's physical activity levels via a bodyweight exercise program and a change in bone density, cognition, and quality of live for patients diagnosed with Multiple Sclerosis. The subjects enrolled in this study will perform a six week training cycle which includes one session per week located at Holy Name Medical Center (physical therapy department) as well as one session per week performed at the subject's home (video guide will be distributed). The training sessions should take approximately 30 minutes and include 3 sets of 10 repetitions for each of the individual exercises. There are five unchanging exercises that will be performed at each training session which include: wall push ups, chair squats, chair dips, step ups, and calf raises. Each subject will be required to perform both training sessions per week for six weeks. The following two weeks are set aside for make up dates for any missed training sessions if needed. During this six to eight week training (treatment) phase, one of the study investigators will remain in contact with the subjects of the study as to ensure commitment of at home training sessions. Prior to the training phase of this study, each subject will have a bone density DEXA scan performed and must complete SDMT (symbol digit modalities test) and MSIS-29 (multiple sclerosis impact scale) evaluations. Both the SDMT and MSIS-29 evaluations with be filled out again within two weeks of the completion of the training phase. 8 weeks after completion of the training phase of the study, each subject will return for a second bone density DEXA scan as well as complete both the SDMT and MSIS-29 evaluations for a third time. The duration of the study will fall between 14 and 16 weeks for any given participant depending on if the additional two weeks are needed to complete the training (treatment) phase. Previous research in this area have supported that bodyweight exercise had a positive impact on fatigue, muscle strength, and balance. Improvements in quality of life as well as cognition have also been documented by MS patients after performing exercise regimen. Because of the positive effects of exercise on patients with MS, the investigators in this study investigated the effects of weight-based training on bone density, cognition, depression, and quality of life in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Diagnosis of RRMS, PPMS, SPMS, or CIS per the 2010 McDonald's criteria [Polman 2011].
* Baseline EDSS score less than 5.5

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Inability to read or understand English.
* Any contraindication to perform weight-based training exercises.
* Use of any supplemental human growth hormone, performance enhancing drug, or anabolic (non-clinical) steroid.
* Participant has become or intends on becoming pregnant.
* Participant has had a relapse in the past 6 months.
* Patients who currently exercise more than three times per week.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Osteopenia | 14 to 16 weeks
  Change in bone density due to the addition of two body weight training sessions per week for a six (to eight) week time period. Bone density will be measured via a DEXA bone density scan at day one of the trial and a secondary DEXA scan taking place eight weeks after the final training session. The duration of this aspect of the study falls between 14 and 16 weeks depending on participant training schedule and if rescheduled or make up training sessions are needed.

SECONDARY OUTCOMES:
Depression and Quality of Life: MSIS (Multiple Sclerosis impact scale) survey/questionnaire | 14 to 16 weeks
  Change in the study participants' view of depression and quality of life pertaining to their MS due to the addition of two body weight training sessions per week for a six (to eight) week time period. Depression and quality of life will be recorded via an (MSIS-29) Multiple Sclerosis Impact Scale survey/questionnaire. This questionnaire consists of 29 items dealing with both the physical and psychological impact of Multiple Sclerosis from a participant's perspective. The MSIS-29 is scored between 29 and 145 in which a higher value indicates a greater impact of MS from a subject's perspective. This questionnaire will be completed by participants on day one of the trial, within two weeks of the completion of their training sessions (between weeks 6 and 10), and eight weeks after their final training session (between weeks 14-16).
Cognition | 14 to 16 weeks
  Change in cognition due to the addition of two body weight training sessions per weeks for a six (to eight) week time period. Cognition will be measured using an SDMT (symbol digit modalities test) on day one of the trial, within two weeks of the completion the final training session (between weeks 6 and 10), and eight weeks after the completion of the final training session (between weeks 14 and 16). The duration of this aspect of the study falls between 14 and 16 weeks depending on participant training schedule and if rescheduled or make up training sessions are needed.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Picone, Principal Investigator — Holy Name Medical Center Multiple Sclerosis Center
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States